CLINICAL TRIAL: NCT06285721
Title: DELirium Treatment With Transcranial Electrical Stimulation
Acronym: DELTES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: A.J.C. Slooter (Other)
Collaborators: Radboud University Medical Center (Other); HagaZiekenhuis (Other)
Responsible Party: Sponsor-Investigator, A.J.C. Slooter, Professor of Intensive Care Neuropsychiatry, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DELTES
Record Dates: First submitted 2024-02-19; First posted 2024-02-29 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Delirium
Keywords: electroencephalography; transcranial alternating current stimulation
MeSH Terms: conditions — Delirium | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standardized treatment arm (Experimental): Standardized tACS will be applied with 2.0 mA (peak-to-peak) intensity for 30 minutes, with a 10 Hz frequency. Two 5x5 cm saline-soaked electrodes located at the frontal and occipito-parietal part of the scalp will be utilized (corresponding to 10-20 EEG electrode locations POz-Oz and AFz), including in the stimulation field the DLPFC, precuneus and posterior cingulate cortex. At the beginning of stimulation, the intensity will ramp up for 30 seconds to 2.0 mA peak-to-peak, while at the end of stimulation, the intensity will ramp down for 30 seconds.
  Interventions: Device: transcranial alternating current stimulation (tACS)
- Personalized treatment arm (Experimental): Personalized tACS will be applied with 2.0 mA (peak-to-peak) intensity for 30 minutes with a 30 second ramp up and ramp down. Treatment will be personalized based on a delirium neural mass model. After fitting the model to the individual EEG, a virtual tACS trial allows for optimization of treatment parameters for each individual patient. Treatment optimization will take place through changing stimulation location and/or frequency. After determining the optimal individual treatment strategy, settings of the personalized stimulation will remain constant during the treatment phase.
  Interventions: Device: transcranial alternating current stimulation (tACS)
- Sham treatment arm (Sham Comparator): At the beginning and end of this 30-minute protocol, the tACS device will ramp up to 2.0 mA peak-to-peak intensity for 30 seconds, stimulate for 60 seconds and ramp down for 30 seconds, which mimics the sensation of actual tACS stimulation and improves blinding.
  Interventions: Device: Sham transcranial alternating current stimulation (tACS)

INTERVENTIONS:
Device: transcranial alternating current stimulation (tACS) — tACS is a non-invasive brain stimulation technique which involves the application of a low intensity electric current between two or more surface electrodes. tACS uses stimulation with a current alternating at a specific frequency that can entrain endogenous neuronal oscillations by inducing neural synchronization. The administration of tACS is proposed to phase-lock large populations of neurons in the superficial layers of the cerebral cortex causing neural synchronization in the corresponding frequency, thereby altering connectivity. tACS will be delivered via a transcranial electrical stimulation (tES) device (Nurostym tES, Brainbox Ltd, United Kingdom). This device has been CE-marked for use as a medical device for the treatment of mental and neurological disorders.
  Arms: Personalized treatment arm; Standardized treatment arm
Device: Sham transcranial alternating current stimulation (tACS) — Sham-tACS is a form of non-effective stimulation which can mimic the subjective sensation of active tACS treatment. During sham-tACS, the device will ramp up to 2.0 mA peak-to-peak intensity for 30 seconds, stimulate for 60 seconds and ramp down for 30 seconds, which mimics the sensation of actual tACS stimulation and improves blinding.The sham-tACS will be delivered via a transcranial electrical stimulation (tES) device (Nurostym tES, Brainbox Ltd, United Kingdom). This device has been CE-marked for use as a medical device for the treatment of mental and neurological disorders.
  Arms: Sham treatment arm

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of standardized and personalized transcranial alternating current stimulation (tACS) in patients with delirium. To investigate this, will perform a double-blind, randomized, sham-controlled, multicenter trial.

To test the safety and feasibility of tACS in delirious patients, the first 30 patients will be randomized to receive either active or sham tACS treatment in a 1:1 ratio through a pilot study. For the main phase of the study, patients will be randomized, resulting in an overall 1:1:1 allocation to standardized tACS, personalized tACS or sham treatment.

Electroencephalogram (EEG) will be measured directly before and directly after the first stimulation session to assess whether tACS can reduce relative delta power. tACS or sham treatment will be given once daily for a maximum of 14 days, or until resolution of delirium or discharge (whichever comes first). During the treatment phase, presence and severity of delirium will be assessed daily. After the treatment phase, an additional EEG will be measured. Cognitive status will be assessed three months after the initial tACS session.

DETAILED DESCRIPTION:
Delirium, a prevalent neuropsychiatric syndrome caused by an underlying medical condition, characterized by cognitive deficits such as inattention, extends hospital stay, increases healthcare costs and increases the risk of long-term cognitive decline. Prolonged and severe delirium is associated with worse long-term outcomes. There is currently no treatment that reduces the duration or severity of delirium.

Delirium is consistently characterized by diffuse oscillatory slowing of the EEG, including pronounced loss of alpha activity and increased relative delta power. Additionally, functional connectivity between brain regions is decreased during delirium. In light of this, tACS is a potential treatment option that directly addresses the brain dysfunction observed in delirium. Because tACS has shown the ability to improve multiple domains of cognition, including attention, and modify functional connectivity, we aim to investigate the effectiveness of tACS as treatment for delirium. We will utilize the EEG to measure the effects of tACS, using relative delta power as a primary outcome measure.

Additionally, EEG measurements can capture individual spectral and connectivity changes targeted with tACS, making EEG a promising input for personalized tACS treatment. Neural mass modelling is a way to model the behavior of groups of neurons resulting in oscillatory output similar to EEG. This type of model is able to represent delirium pathology and, when combined with individual EEG input, can be employed to optimize treatment effectiveness, leading to personalized tACS treatment.

The overarching aim of the study is to investigate whether treatment with tACS, either standardized or personalized, induces EEG alterations indicative of reversal of delirium. The primary outcome is relative delta power in the EEG measured after the first tACS session. Secondary outcomes include severity and/or duration of delirium measured with validated delirium assessment instruments.

Patients aged 50 years and older with delirium that persists for at least 2 days, despite adequate treatment of underlying causes will be included in the study (n = 159). Inclusion will take place in the intensive care unit (ICU) and non-ICU wards of the University Medical Centre (UMC) Utrecht, Radboud UMC and HagaZiekenhuis.The proposed tACS protocol is considered safe according to the latest published international safety guidelines. All participants will be screened for their relevant medical history and other tACS safety aspects.

ELIGIBILITY:
Inclusion Criteria:

* Age over 50 years.
* Diagnosis of delirium
* Richmond Agitation and Sedation Scale (RASS) score of -2 to +2.
* Delirium duration of at least two days prior to study inclusion, based delirium assessments and/or descriptions in the medical and/or nursing files.
* Known causes underlying delirium are being treated adequately, as assessed by the treating physician.

Exclusion Criteria:

* Inability to conduct delirium assessment (e.g. coma, deaf, blind) or inability to speak Dutch or English.
* A moribund state.
* Alcohol/substance abuse withdrawal or stroke as precipitating factor for delirium.
* Diagnosis of dementia, based on medical record review and/or a score of ≥4.5 on the short form of the Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE)
* One or more contra-indications for tACS:

  1. History of serious head trauma or brain surgery;
  2. Large or ferromagnetic metal parts in the head (except for a dental wire);
  3. Implanted cardiac pacemaker or neurostimulator;
  4. Skin diseases or inflammations;
  5. Epilepsy.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Relative delta power | 1 day
  Calculated by dividing the absolute power in the delta frequency range by the total power, assessed using 64-channel resting-state EEG directly before and after tACS.

SECONDARY OUTCOMES:
Duration of delirium | Two weeks
  Delirium duration is evaluated by counting the number of days delirium is observed during the treatment period. We utilize the Intensive Care Delirium Screening Checklist (ICDSC), comprising 8 items, with a score of 4 or higher indicating the presence of delirium. Additionally, the Richmond Agitation-Sedation Scale (RASS), a 10-point scale ranging from +4 to -5, is used to assess the level of sedation (-5 indicating total sedation, +4 indicating combative behavior). A RASS score of -4 or lower, followed by an ICDSC score of 4 or higher, is also considered a delirium day.
Severity of delirium | Two weeks
  The cumulative score on the Intensive Care Delirium Screening Checklist (ICDSC), which includes 8 items and has a score range of 0-8, is documented for each day where delirium is observed during the hospital admission. In instances where the ICDSC score is unavailable, it will be approximated using information retrieved from the electronic patient record and standard delirium assessment tools routinely conducted.
Length of hospital stay | 3 months
  The total number of days admitted to hospital
Cognitive status three months post delirium | 3 months
  Score on the Telephone Interview for Cognitive Status Modified (TICS-M). The TICS-M is a brief, 13-item test of cognitive functioning with scores ranging from 0 to 50, with higher scores indicating better cognitive performance.
Subjective sensations during treatment | Two weeks
  Score on three-point Likert-type scale to assess sensations experienced during transcranial alternating current stimulation (tACS). The scale ranged from 0, indicating 'no sensation,' to 1, indicating 'slight sensation,' and 2, indicating 'intense sensation.' These sensations included itch, pain, burning sensation, heat, iron taste, headache, neck pain, phosphenes, dizziness, and nausea.
Average peak frequency | Two weeks
  Average peak frequency values will be calculated by averaging, over epochs, the peak frequency, assessed using 64-channel resting-state EEG before and after tACS and during the follow-up measurement.
Phase Lag Index | Two weeks
  Phase lag index captures phase synchronization between different EEG channels, assessed using 64-channel resting-state EEG before and after tACS and during the follow-up measurement.
Corrected Amplitude Envelope Correlation (AECc) | Two weeks
  AECc captures amplitude synchronization between different EEG channels, assessed using 64-channel resting-state EEG before and after tACS and during the follow-up measurement.
Relative power | Two weeks
  Relative power will be calculated by dividing the absolute power of the frequency band by the total absolute power in the EEG, assessed using 64-channel resting-state EEG before and after tACS and during the follow-up measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Arjen JC Slooter, MD, PhD, Principal Investigator — UMC Utrecht
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - HagaZiekenhuis, The Hague, South Holland

IPD SHARING:
Plan to Share IPD: Yes
Patients can specify whether they agree to share their data with other research institutes. Depending on consent of participants, we might be able to share IPD after publication of results.
Time Frame: After first published results, no end date
Access Criteria: After approval of the consortium members

REFERENCES:
- [Derived] van der A J, Lodema Y, Ottens TH, Schutter DJLG, Emmelot-Vonk MH, de Haan W, van Dellen E, Tendolkar I, Slooter AJC. DELirium treatment with Transcranial Electrical Stimulation (DELTES): study protocol for a multicentre, randomised, double-blind, sham-controlled trial. BMJ Open. 2024 Nov 2;14(11):e092165. doi: 10.1136/bmjopen-2024-092165. PMID 39488424